CLINICAL TRIAL: NCT00737490
Title: Does Echocardiographically Guided Ventriculo-Ventricular Optimization Yield a Sustained Improvement in Echocardiographic Parameters in Cardiac Resynchronization Therapy Patients? (DEVISE CRT)
Acronym: Devise-CRT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: Pro00007865; 7314
Record Dates: First submitted 2008-05-04; First posted 2008-08-19 (Estimated); Last update posted 2014-08-01 (Estimated); Status verified 2013-04

CONDITIONS: Cardiomyopathy; Heart Failure
MeSH Terms: conditions — Cardiomyopathies; Heart Failure

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Echocardiographically guided optimized device programming: specifically sequential BiV pacing. "Sequential Arm"
  Interventions: Other: "Sequential Arm" (Promote , model # 2207-36 or Atlas HF , model # V-343)
- 2 (Active Comparator): Simultaneous BiV pacing. "Simultaneous Arm"
  Interventions: Other: "Simultaneous Arm" (Promote , model # 2207-36 or Atlas HF , model # V-343)

INTERVENTIONS:
Other: "Sequential Arm" (Promote , model # 2207-36 or Atlas HF , model # V-343) — Echocardiographically guided optimized device programming: specifically sequential BiV pacing. "Sequential Arm"
  Using one of the FDA approved St. Jude devices, depending on MD preference.
  Arms: 1
Other: "Simultaneous Arm" (Promote , model # 2207-36 or Atlas HF , model # V-343) — simultaneous BiV pacing.
  Using one of the FDA approved St. Jude devices, depending on MD preference.
  Arms: 2

SUMMARY:
The purpose of this study is to determine whether using an echocardiogram (a painless test where ultrasound is used to see your heart) while using mild electrical stimulation from your own CRT-D device to stimulate the ventricles (the lower chambers of the heart) to squeeze one slightly earlier than the other will show a sustained increase your heart's productivity (Cardiac Output (CO)), following implantation of a Cardiac Resynchronization Device (CRT-D). We believe that squeezing some parts of the heart earlier than others may make the heart a stronger pump.

ELIGIBILITY:
Inclusion Criteria:

1. LVEF </= 35% as assessed by echocardiography.
2. New York Heart Association Functional Class III or IV CHF despite contemporary medical therapy for CHF.
3. QRS duration of >/= 120 ms.
4. Ability to provide written, informed consent.
5. Age > 18 years.
6. Successful implant of a biventricular/ICD pacemaker device.

Exclusion Criteria:

1. Documented Chronic Atrial Fibrillation
2. Life expectancy less that 6 months due to non-cardiac causes
3. Inability to place a coronary sinus left ventricular pacing lead
4. Pregnancy
5. Scheduled cardiac surgery within the next 6 months
6. Prosthetic Tricuspid Valve

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2005-06; Primary Completion 2009-12 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
To determine if a sustained hemodynamic benefit of increased Cardiac Output is maintained in patients who undergo ECHO guided optimization of V-V timing following CRT implantation when compared to patients simultaneously biventricularly paced. | 6 months

SECONDARY OUTCOMES:
Assessment for improvements in 1)6 minute walk 2)ECHO parameters 3)symptoms as assessed by the Minnesota Quality of Life Score. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Hranitzky Patrick, MD, Principal Investigator — Duke University; Patrick Hranitzky, MD, Study Director — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States